CLINICAL TRIAL: NCT00053807
Title: Adjuvant Interleukin-2, Interferon-alpha and 5-Fluorouracil for Patients With High Risk of Relapse After Surgical Treatment for Renal Cell Carcinoma
Brief Title: Interleukin-2, Interferon Alfa, and Fluorouracil Compared With Observation in Treating Patients Who Have Undergone Surgery for Kidney Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-30955; EORTC-30955
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Kidney Cancer
Keywords: stage III renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — aldesleukin; Interferon-alpha; Fluorouracil; Chemotherapy, Adjuvant

INTERVENTIONS:
Biological: aldesleukin
Biological: recombinant interferon alfa
Drug: fluorouracil
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of tumor cells. Interleukin-2 may stimulate a person's white blood cells to kill tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining interferon alfa and interleukin-2 with fluorouracil may kill any remaining tumor cells following surgery. It is not yet known whether combining interferon alfa and interleukin-2 with fluorouracil is more effective than observation after surgery for kidney cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of combining interleukin-2, interferon alfa, and fluorouracil to that of observation alone in treating patients who have undergone surgery for kidney cancer and are at high risk of relapse.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effect of adjuvant combination therapy comprising interleukin-2, interferon alfa, and fluorouracil vs observation only on disease-free survival or overall survival of patients with renal cell carcinoma at high risk of relapse after radical surgery.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive interleukin-2 subcutaneously (SC) on days 3, 4, and 5 of weeks 1 and 4 and on days 1, 3, and 5 of weeks 2 and 3. Patients also receive interferon alfa SC once weekly during weeks 1 and 4 and 3 times weekly during weeks 2, 3, 5, 6, 7, and 8. Patients then receive fluorouracil IV on day 1 of weeks 5, 6, 7, and 8.
* Arm II (control arm): Patients receive no adjuvant treatment before disease progression.

Quality of life is assessed at baseline and at 2 and 6 months after randomization.

Patients are followed monthly for 3 months (arm I only), every 3 months for 1 year, every 6 months for 4 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 550 patients (275 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary renal cell carcinoma meeting 1 of the following criteria:

  * Stage T3b, T3c, or T4 tumor
  * Any pT stage and nodal status pN 1 or 2
  * Any pT stage and microscopic positive margins
  * Presence of any microscopic vascular invasion
* Underwent surgical resection of primary tumor within the past month

  * Removal of clinical N+ disease required
* No evidence of metastatic disease
* No evidence of macroscopic residual disease

PATIENT CHARACTERISTICS:

Age

* 75 and under

Performance status

* WHO 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Liver function tests no greater than 1.25 times upper limit of normal (ULN)

Renal

* Creatinine less than 1.5 times ULN

Cardiovascular

* No myocardial infarction within the past 6 months
* No unstable angina pectoris

Other

* Not pregnant or nursing
* No prior or other concurrent malignancies that would preclude study therapy or comparisons
* No other concurrent illness that would preclude study therapy
* No concurrent active infections requiring antibiotic therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No other concurrent immunotherapy

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* No concurrent corticosteroids
* No concurrent hormonal therapy

Radiotherapy

* No prior radiotherapy

Surgery

* See Disease Characteristics
* No prior major organ allografts

Other

* No other concurrent investigational drugs, agents, or devices

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 1998-02; Primary Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pieter H. M. de Mulder, MD, PhD, Study Chair — Universitair Medisch Centrum St. Radboud - Nijmegen; Hein van Poppel, MD, PhD, Study Chair — University Hospital, Gasthuisberg; Paul A. Vasey, MD, Study Chair — Beatson Institute for Cancer Research - Glasgow
Locations (17):
- Kaiser Franz Josef Hospital, Vienna, Austria
- Belgium (4):
  - Onze Lieve Vrouw Ziekenhuis Aalst, Aalst
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Groeninge - Campus St. Maarten, Kortrijk
  - U.Z. Gasthuisberg, Leuven
- National Institute of Oncology, Budapest, Hungary
- Rambam Medical Center, Haifa, Israel
- Ospedale di Circolo e Fondazione Macchi, Varese, Italy
- Netherlands (6):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Akademisch Medisch Centrum, Amsterdam
  - University Medical Center Nijmegen, Nijmegen
  - Daniel Den Hoed Cancer Center at Erasmus University Medical Center, Rotterdam
  - Academisch Ziekenhuis Utrecht, Utrecht
- Turkey (Türkiye) (2):
  - Marmara University Hospital, Istanbul
  - Dokuz Eylul University School of Medicine, Izmir
- Beatson Institute for Cancer Research - Glasgow, Glasgow, Scotland, United Kingdom

REFERENCES:
- [Result] Aitchison M, Bray CA, Van Poppel H, et al.: Final results from an EORTC (GU Group)/NCRI randomized phase III trial of adjuvant interleukin-2, interferon alpha, and 5-fluorouracil in patients with a high risk of relapse after nephrectomy for renal cell carcinoma (RCC). [Abstract] J Clin Oncol 29 (Suppl 15): A-4505, 2011.